CLINICAL TRIAL: NCT02432547
Title: A Phase IV Randomised Clinical Trial of Laser Therapy for Peripheral Retinal Ischaemia Combined With Intravitreal Aflibercept (Eylea®) Versus Intravitreal Aflibercept Monotherapy for Diabetic Macular Oedema
Brief Title: Laser Therapy Combined With Intravitreal Aflibercept vs Intravitreal Aflibercept Monotherapy (LADAMO)
Acronym: LADAMO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sydney (Other)
Collaborators: Center for Eye Research Australia (Other)
Responsible Party: Principal Investigator, Mark Gillies, Head of Macular Research Group, University of Sydney
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: X14-0157
Record Dates: First submitted 2015-04-23; First posted 2015-05-04 (Estimated); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Diabetic Retinopathy
Keywords: Diabetic; Macular Oedema; Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy; Macular Edema; Retinal Diseases | interventions — aflibercept; Lasers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aflibercept Monotherapy (Active Comparator): Intravitreal aflibercept injections according to a treat and extend regimen.
  Interventions: Drug: Aflibercept
- Targeted laser therapy with Aflibercept (Experimental): Targeted laser photocoagulation therapy to areas of peripheral retinal ischaemia and intravitreal aflibercept injections using a treat and extend regimen.
  Interventions: Drug: Aflibercept; Procedure: Targeted laser therapy

INTERVENTIONS:
Drug: Aflibercept — Aflibercept is a soluble decoy receptor and is produced by fusing all-human DNA sequences of the second immunoglobulin (Ig) domain of human VEGF receptor (VEGFR) 1 to the third Ig domain of human VEGFR-2, which are then fused to the Fc region of human IgG-1. By binding to VEGF-A, aflibercept prevents activation of the native VEGF receptors, VEGFR-1 and VEGFR-2. The study sites will be supplied by Bayer with aflibercept. Intravitreal injection of 2mg in 0.05 ml aflibercept will be administered to the study eye, according to a pre-defined treat and extend regimen.
  Other Names: Eylea
Procedure: Targeted laser therapy — In the experimental group, targeted laser photocoagulation will be applied to areas of peripheral retinal ischaemia 1 month after the initial intravitreal aflibercept. The trial design allows another session of targeted laser photocoagulation 1 month later to complete the treatment if required. Wide-field photography is planned at 3 months to determine if further targeted laser photocoagulation is required, and if so a third session can be applied. The laser settings are based on those used in current clinical practice and have been prospectively defined in the protocol.
  Other Names: Laser
  Arms: Targeted laser therapy with Aflibercept

SUMMARY:
This will be a 24 month phase IV, randomised, prospective, multicentre, clinical trial of laser therapy to areas of peripheral retinal ischaemia combined with intravitreal aflibercept versus intravitreal aflibercept monotherapy. Both arms will have 2mg intravitreal aflibercept according to a treat and extend protocol.

The specific aim of the study is to test whether laser therapy of peripheral retinal ischaemia reduces the overall number of intravitreal aflibercept injections required to control DMO over a 24 month period.

DETAILED DESCRIPTION:
Diabetic retinopathy is the most common cause of blindness in individuals between the ages of 20 and 65 years in developed countries. Swelling of the central retina, or "macular oedema", is the commonest cause of visual loss in diabetic retinopathy.

Recent studies have suggested peripheral retinal ischaemia contributes to macula oedema in diabetes and retinal vein occlusions. Intravitreal anti-Vascular Endothelial Growth Factor (VEGF) therapy, such as Aflibercept (Eylea) has shown encouraging results in managing Diabetic Macular Oedema (DMO). There is evidence that regular treatment with anti-VEGF drugs reduces DMO and improves vision on average.

Previous research at this institution has shown that an average of between 7 and 11 injections are required in the first year to stabilise the disease. However, there is a significant burden to patients in terms of frequent visits to the eye specialist, time off work and repeated injections into the eye. The purpose of this study is to see whether targeted peripheral retinal laser therapy to areas of the retina with impaired blood supply can reduce the number of intravitreal aflibercept injections required over 2 years to stabilise DMO.

ELIGIBILITY:
Inclusion Criteria:

* At screening, the study eye must have DMO with retinal thickness > 300 microns in central 1mm subfield on Spectral domain OCT
* Age >= 18 years
* Diagnosis of diabetes mellitus
* Best corrected visual acuity of 35-79 LogMAR letters at 4 meters (approximately 6/7.5-6/60) in the study eye
* Women of childbearing potential must have a negative urine pregnancy test at the screening visit and prior to treatment. A woman is considered of childbearing potential unless she is postmenopausal and without menses for 12 months or is surgically sterilised
* Peripheral retinal ischaemia affecting an area greater than 10 disc diameters of the wide-field fundus fluorescein angiogram (as per the Central Vein Occlusion Study)
* Centre involving DMO, which in the opinion of the investigator, would not benefit from focal macular laser treatment (e.g. diffuse leak from the capillary bed, disruption of the foveal avascular zone or perifoveal capillary dropout, complete macular grid laser).
* Written informed consent has been obtained

Exclusion Criteria:

* Known allergy to aflibercept or agents used in the study
* Women who are pregnant, nursing, or planning a pregnancy, or who are of childbearing potential and not using reliable means of contraception
* Loss of vision due to other causes (e.g. age related macular degeneration, myopic macular degeneration, retinal vein occlusion) in the study eye.
* Macular oedema due to other causes in the study eye.
* Macula hole, vitreo-macular traction or significant epiretinal membrane in the study eye.
* An ocular condition that would prevent visual acuity improvement despite resolution of oedema (such as foveal atrophy or substantial premacular fibrosis)
* Treatment with intravitreal triamcinolone acetonide (IVTA) within the last 6 months or peribulbar triamcinolone within the last 3 months, or anti-VEGF drugs (bevacizumab, ranibizumab or aflibercept) within the last 2 months in the study eye.
* Cataract surgery within the last 3 months in the study eye
* Previous PRP laser treatment in the study eye
* Previous vitrectomy in study eye
* Media opacity including cataract that already precludes adequate macular photography or cataract that is likely to require surgery within 12 months
* Intercurrent severe disease such as septicaemia, any condition which would affect follow-up or photographic documentation (e.g. geographical, psycho-social)
* History of chronic renal failure requiring dialysis or renal transplant
* Blood pressure >180/110
* Patient has a condition or is in a situation that in the investigator's opinion may put the patient at significant risk, may confound the study results, or may interfere significantly with the patient's participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2022-05-24 (Actual); Study Completion 2022-05-24 (Actual)

PRIMARY OUTCOMES:
Number of intravitreal aflibercept injections over 24 months | 24 months
  Number of intravitreal aflibercept injections in each of the 2 groups required over 24 months

SECONDARY OUTCOMES:
Number of intravitreal aflibercept injections over 12 months | 12 months
  Number of intravitreal aflibercept injections in each of the 2 groups required over 12 months
Proportion of eyes that have central macular thickness <300 microns at 12 months | 12 months
Mean change in central macular thickness (CMT) as measured by OCT at 12 months | 12 months
Mean change in best corrected visual acuity | 12 months
  Mean change in best corrected visual acuity at 12 months
Any change in best corrected visual acuity at 12 months | 12 months
  Any change in best corrected visual acuity at 12 months
Effect of peripheral retinal ischaemia on number of aflibercept injections | 12 months
  Correlation between area of peripheral retinal ischaemia and number of intravitreal injections required at 12 months
Disc vessel measurement | 12 months
  Change in disc vessel diameter at 12 months
Number of intravitreal aflibercept injections in each of the 2 groups required over 24 months | 24 months
Proportion of eyes that have central macular thickness <300 microns at 24 months | 24 months
Mean change in central macular thickness (CMT) as measured by OCT at 24 months | 24 months
Mean change in best corrected visual acuity | 24 months
  Mean change in best corrected visual acuity at 24 months
Any change in best corrected visual acuity at 24 months | 24 months
  Any change in best corrected visual acuity at 24 months
Effect of peripheral retinal ischaemia on number of aflibercept injections | 24 months
  Correlation between area of peripheral retinal ischaemia and number of intravitreal injections required at 24 months
Disc vessel measurement | 24 months
  Change in disc vessel diameter at 24 months
Time until vision stabilisation | 24 months
  Length of time from baseline to vision stabilisation
Quality of life assessment | 24 months
  Quality of life assessment using IVI and NEI VFQ-25 forms at 24 months
Change in area of macular hard exudates | 24 months
  Change in area of macular hard exudates from baseline to 24 months
Change in distance of closest hard exudate from the foveal centre | 24 months
  Change in distance of closest hard exudate from the foveal centre between baseline and 24 months
Mean change in treatment interval over time | 24 months
  Mean change in treatment interval between intravitreal aflibercept injections over time

OTHER OUTCOMES:
Mean change in foveal avascular zone | 24 months
  Mean change in maximum diameter of foveal avascular zone at 24 months
Incidence of requirement for rescue macular laser treatment | 24 months
  Incidence of requirement for rescue macular laser treatment
Ocular adverse events | 24 months
  Incidence and severity of ocular adverse events including severe (>15 letter) loss of vision
Non-ocular adverse events | 24 months
  Incidence and severity of non-ocular adverse events
Change in visual field from baseline | 24 months
  Incidence of new visual field defect that would fail to meet driving standard at 24 months. (Selected study sites only).
Development of new neovascular complexes on posterior pole OCT imaging | 24 months
  Incidence of new neovascular complexes at 24 months
Development of new proliferative diabetic retinopathy on wide-field fluorescein angiography | 24 months
  Incidence of new proliferative diabetic retinopathy at 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Samantha Fraser-Bell, PhD FRANZCO, Principal Investigator — Save Sight Institute
Locations (2):
- Australia (2):
  - Save Sight Institute, Sydney, New South Wales
  - Centre for Eye Research Australia, Melbourne, Victoria